CLINICAL TRIAL: NCT06472713
Title: A Prospective, Single-arm Phase 2 Study Evaluating the Efficacy and Safety of Mitoxantrone Hydrochloride Liposome Injection Combined with PD-1 Blockade in Previously Treated Recurrent or Metastatic Nasopharyngeal Carcinoma
Brief Title: Clinical Study of Mitoxantrone Hydrochloride Liposome Combined with PD-1 Blockade in Recurrent or Metastatic NPC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ming-Yuan Chen (Other)
Responsible Party: Sponsor-Investigator, Ming-Yuan Chen, Archiater, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZDWY.BYAFZZX.027
Record Dates: First submitted 2024-06-15; First posted 2024-06-25 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-06

CONDITIONS: Recurrent or Metastatic Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; Recurrent; Metastatic; Mitoxantrone Hydrochloride Liposome; PD-1 Blockade
MeSH Terms: conditions — Recurrence; Nasopharyngeal Carcinoma; Neoplasm Metastasis | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mitoxantrone group (Experimental): Mitoxantrone hydrochloride liposome (30 mg/cycle) injection combined with PD-1 blockade (comprising tislelizumab <200 mg/cycle>, carrellimab <200 mg/cycle>, or toripalimab <240 mg/cycle>) once every 3 weeks for up to 8 cycles, following the uniform PD-1 blockade alone once every 3 weeks for two years, or until intolerable toxicity, subject withdrawal of informed consent, initiation of new antitumor therapy, loss of follow-up, or death, whichever occurs first.
  Interventions: Drug: Mitoxantrone hydrochloride liposome injection; Drug: PD-1 Inhibitors

INTERVENTIONS:
Drug: Mitoxantrone hydrochloride liposome injection — Mitoxantrone hydrochloride liposome injection once every 3 weeks for up to 8 cycles or until intolerable toxicity, subject withdrawal of informed consent, diseases progression, initiation of new antitumor therapy, loss of follow-up, or death, whichever occurs first.
Drug: PD-1 Inhibitors — PD-1 blockade (comprising tislelizumab <200 mg/cycle>, carrellimab <200 mg/cycle>, or toripalimab <240 mg/cycle>) once every 3 weeks for two years, or until intolerable toxicity, subject withdrawal of informed consent, diseases progression, initiation of new antitumor therapy, loss of follow-up, or death, whichever occurs first.

SUMMARY:
This is a prospective, single-arm Phase 2 study to evaluate the efficacy and safety of mitoxantrone hydrochloride liposome injection combined with PD-1 blockade in patients with recurrent (not unable to locally curative treatment) or metastatic NPC who failed at least first-line platinum-containing standard regimen and/or anti PD-1/L1.

DETAILED DESCRIPTION:
Thirty-two recurrent (not unable to locally curative treatment) or metastatic NPC patients who had failed at least first-line platinum-containing standard regimen and/or anti PD-1/L1 were eligible to receive mitoxantrone hydrochloride liposome injection combined with PD-1 blockade once every 3 weeks for up to 8 cycles, following PD-1 blockade alone once every 3 weeks for 2 years. All patients will be treated until disease progression as determined by the investigator based on RECIST 1.1 criteria, intolerable toxicity, subject withdrawal of informed consent, initiation of new antitumor therapy, loss of follow-up, death, or study completion, whichever occurs first. Regular visits and imaging examinations will be conducted to evaluate the efficacy and safety of the treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate in the study, sign the informed consent form (ICF), and comply with study plan visits, treatment plans, laboratory tests, and other study procedures.
2. Nasopharyngeal carcinoma confirmed by histopathology (differentiated or undifferentiated non-keratinous carcinoma).
3. Age ≥ 18 & ≤ 70 years.
4. PS (Performance Status) score 0-1.
5. Recurrent or metastatic nasopharyngeal carcinoma that has failed first-line platinum-containing standard regimen and/or second-line standard regimen failure.
6. Previously received at least one line of systemic therapy. (Progression after radical concurrent chemoradiotherapy, during neoadjuvant or adjuvant therapy, or within 6 months after the end of treatment can be recorded as 1-line therapy).
7. Recurrent or metastatic nasopharyngeal carcinoma that has failed anti PD-1/L1: anti PD-1/L1 exposure at least 6 weeks, and the protocol used at the time of enrollment in this study meets one of the following two points: (1) Relapse during adjuvant therapy after radiotherapy, or relapse within 6 months after the end of treatment; (2) First-line treatment phase, progression during anti PD-1/L1 treatment, or progression within 3 months after the end of anti PD-1/L1 (whether combined with chemotherapy/targeting drugs);
8. At least one measurable lesion according to RECIST 1.1 criteria (the spiral CT scan diameter of the measurable lesion is ≥ 10 mm or the short diameter of the enlarged lymph node is ≥15mm ); lesions that have undergone local treatment can be selected as target lesions if there is clear evidence of significant progress compared to the end of treatment.
9. All acute toxicities of previous antitumor therapy have returned to ≤ grade 1 (according to NCI-CTCAE v5.0) or reached the level specified in the inclusion/exclusion criteria. (Except for partial toxicity, such as alopecia, hair color change, nail change, fatigue, etc., which do not pose safety risks to subjects).
10. Adequate main organ function. a. Hematology: neutrophil absolute value (ANC) ≥1.5×10^9/L, hemoglobin (Hb) ≥ 9.0 g/dL, platelets ≥ 100×10^9/L; b. Liver function: bilirubin ≤ 1.5 times the upper limit of normal (ULN) (patients with known Gilbert disease and serum bilirubin level ≤ 3 times ULN could be enrolled; patients with liver metastasis, ≤ 5 times ULN), AST and ALT ≤ 3 times ULN, and alkaline phosphatase ≤ 3 times ULN; Albumin ≥ 3 g/dL; c. International Normalized ratio (INR) or prothrombin time (PT) or activated partial thromboplastin time (aPTT) ≤ 1.5 times; d. Renal function: serum creatinine ≤ 1.5 ULN or creatinine clearance ≥ 60 mL/min according to Cockcroft-Gault formula; e. Proteinuria: urinary protein/creatinine ratio (UPC ratio) < 1.0. If the UPC ratio is less than or equal to 0.5, no further check is required. Patients with UPC ratio > 0.5 and those with 24-hour urinary protein < 1000 mg could be enrolled; f. Note: The UPC ratio of random urine is a quantitative estimate of 24-hour urinary protein, and the two have a good correlation. UPC ratio can be calculated using the following formula: (a) Urinary protein/urinary creatinine (if both protein and creatinine are mg/dL); (b) (urinary protein)*0.088/ urinary creatinine (if urinary creatinine is mmol/L).
11. Survival is expected to be ≥ 3 months.
12. Female subjects with negative blood human chorionic gonadotropin (HCG) (except for menopause and hysterectomy), female subjects of reproductive age and their partners using effective contraception during the trial period and within 6 months after the end of the last dose (e.g. Combined hormones [containing estrogen and progesterone combined to inhibit ovulation, progesterone contraception combined to inhibit ovulation, IUD, intrauterine hormone release system, bilateral tubal ligation, vasectomy, abstinence from sex, etc.).
13. Male patients and their partners agree to use one of the contraceptive measures described in Article 9.

Exclusion Criteria:

1. Recurrent lesions in local areas suitable for radical method (surgery) treatment.
2. Severe allergy to mitoxantrone or liposome (such as systemic rash/erythema hypotension, bronchospasm, angioedema, or anaphylaxis).
3. Prior treatment with doxorubicin or other anthracyclines and the cumulative doxorubicin doses greater than 350 mg/m^2 (anthracycline equivalent: 1 mg doxorubicin = 2 mg epirubicin = 2 mg daunorubicin = 0.5 mg normethoxydaunorubicin = 0.45 mg mitoxantrone).
4. Estimated survival < 3 months.
5. Diagnosed and/or treated with other malignancies within 5 years prior to initial administration. (except for cervical cancer, skin basal cell or squamous cell carcinoma, localized prostate cancer, and ductal carcinoma in situ after radical treatment).
6. Received surgery, chemotherapy, radiotherapy, immunotherapy, or any investigational drug or other antitumor therapy within the 4 weeks prior to initial administration (less than 2 weeks after palliative radiotherapy).
7. Patients with hypertension who cannot be reduced to the normal range by antihypertensive drugs (systolic blood pressure > 140 mmHg/ diastolic blood pressure > 90 mmHg); Have ≥ grade II coronary heart disease; Any of the following conditions occurred during the first 6 months of enrollment: Myocardial infarction, severe/unstable angina pectoris, NYHAII grade or higher cardiac insufficiency, grade 2 or higher persistent arrhythmias (including prolonged QTc interval > 450ms in men), Women > 470ms), any grade of atrial fibrillation, coronary/peripheral artery bypass grafting, symptomatic congestive heart failure, or cerebrovascular accident (including transient ischemic attack or symptomatic pulmonary embolism); The ejection fraction of the heart is below 50% or below the lower limit of the range of laboratory tests at the study center. Patients with a history of arterial thromboembolism events and venous thromboembolism > grade 3. (Patients with S-T elevation ≥ 2mm on the ECG may be enrolled if they do not show signs of recent myocardial infarction or ischemia) (according to NCI-CTCAE v5.0).
8. Severe infection (such as intravenous antibiotics, antifungals, or antivirals as required by clinical practice) during the 4 weeks prior to the first dose, or any unexplained fever >38.5 ° C during the screening period / 7 days prior to the first dose, or white blood cell count >15×109/L at baseline.
9. Immunosuppressants, or systemic hormone therapy (dose >10mg/ day of prednisone or other therapeutic hormone) are being used for the purpose and continue to be used within 2 weeks before the first dose.
10. The subject has any active autoimmune disease or history of autoimmune disease (including but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, pituitaritis, nephritis, hyperthyroidism, hypothyroidism; Patients with vitiligo or who had complete remission of asthma in childhood and did not require any intervention as adults were included; Patients with asthma requiring medical intervention with bronchodilators were not included).
11. Exacerbations of COPD or other respiratory diseases requiring hospitalization within 1 month prior to registration.Patients with active tuberculosis (TB) who are receiving anti-TB therapy or have received anti-TB therapy within 1 year prior to screening.
12. HIV-positive people; HBsAg positive and HBV DNA copy number positive (quantitative detection ≥1000 cps/ml); Chronic hepatitis C blood screening positive (HCV antibody positive).
13. Live vaccine was administered within 4 weeks before the first dose or possibly during the study period.
14. Pregnant or lactating women.
15. Women with reproductive potential and sexually active men who are unwilling/unable to use medically acceptable forms of contraception.
16. Have any serious and/or uncontrollable medical conditions that, as determined by the investigator, may affect the patient's participation in the study, such as alcoholism, drug abuse, other serious diseases (including mental illness) that require combined treatment, serious laboratory abnormalities, and family or social factors that affect the safety of the patient.
17. Other situations that the investigator determines to be inappropriate for participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-07-20 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Through study completion, an average of 2 years
  Objective response rate (ORR) is defined as the proportion of patients with a complete response or partial response to treatment

SECONDARY OUTCOMES:
Duration of Response (DOR) | Through study completion, an average of 2 years
  Duration of Response (DOR) is defined as time from the first assessment of CR or PR until the date of the first occurrence of PD, or until the date of death
Disease control rate (DCR) | Through study completion, an average of 2 years
  Disease Control Rate (DCR) is defined as the percentage of patients who have achieved complete response, partial response and stable disease to a therapeutic intervention in clinical trials of anticancer agents
Progression-free survival (PFS) | Through study completion, an average of 2 years
  Progression-Free Survival PFS is defined as the time from randomization to progression or death
Overall survival (OS) | Through study completion, an average of 2 years
  Overall survival (OS) is defined as the duration from the date of diagnosis to death or last follow-up, with no restriction on the cause of death.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Affiliated Hospital, Sun Yat-sen University, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Data can be requested from the corresponding author beginning 1 year after publication of the study.